CLINICAL TRIAL: NCT05212545
Title: Randomised Double-blind 4-arm Parallel, Placebo-controlled Trial Investigating the Effects of Prebiotics Alone or in a Combination on Intestinal Colonization and Ability to Influence Mood in a University Cohort
Brief Title: Effects of Prebiotics on Intestinal Colonization and Mood in a University Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21017m-jhr
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Mood

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 10 g maltodextrin per day
  Interventions: Dietary Supplement: Placebo
- Prebiotic Supplement (Experimental): 10 g Prebiotic supplement + maltodextrin per day
  Interventions: Dietary Supplement: Prebiotic supplement
- Prebiotic combination (Experimental): 10 g prebiotic supplement+ prebiotic oligosaccharide per day
  Interventions: Dietary Supplement: Prebiotic combination
- prebiotic oligosaccharide (Experimental): 10 g maltodextrin + prebiotic oligosaccharide per day
  Interventions: Dietary Supplement: Prebiotic oligosaccharides

INTERVENTIONS:
Dietary Supplement: Placebo — maltodextrin taken daily for 4 weeks with water
  Arms: Placebo
Dietary Supplement: Prebiotic supplement — Prebiotic supplement taken daily for 4 weeks with water
  Arms: Prebiotic Supplement
Dietary Supplement: Prebiotic combination — prebiotic oligosaccharides mixture taken daily for 4 weeks with water
  Arms: Prebiotic combination
Dietary Supplement: Prebiotic oligosaccharides — Prebiotic oligosaccharides taken daily for 4 weeks with water
  Arms: prebiotic oligosaccharide

SUMMARY:
There is a growing interest within the scientific community of whether prebiotics can aid in clinical outcomes including mood via modulation of the gut microbiota and its resulting metabolites via the gut-brain axis. This is especially prevalent given that mental health conditions are associated with cost and burden on the health care system. Yet, to date very few studies have investigated the potential effects of prebiotics to influence mood via the modulation of the gut microbiota with previous studies recording mixed results indicating further work in this area would be highly beneficial.

DETAILED DESCRIPTION:
Several reports have suggested that poor mental health among university students is on the increase. Factors driving this; including academic pressure, overdemanding workloads, financial concerns, and peer pressure; can adversely affect academic performance and self-worth. Thus, there is an increasing need to develop new strategies to help tackle these modalities while also reducing the burden on the health system.

In recent years there has been increasing interest in the bi-directional relationship that exists between the gut and the brain, a term coined the gut-brain axis, and it is suggested to play a role in influencing mood via chemical messengers.

As diet is key manipulator of the gut microbiota one way to influence the composition of the gut is via diet and the use of functional foods including prebiotic oligosaccharides.

The idea that functional foods like prebiotics may help to affect mood holds particular appeal due to them being relatively free of side effects, cheap, readily accessible and possessing additional health benefits including improving bowel transit function and improving satiety amongst others. Yet, to date previous research on the potential for prebiotics has produced mixed results due to differences in the populations tested, doses and types of prebiotics used, and means of assessing changes in mood suggesting further work in this area would be highly beneficial.

Therefore, this present study aims to address the question "can manipulation of the gut microbiota using prebiotic oligosaccharides alone or in combination influence mental state in a taught university student population?".

ELIGIBILITY:
Inclusion Criteria:

* Volunteer is healthy at the time of pre-examination
* Possess mild/moderately elevated levels of stress
* Volunteer is aged ≥ 18 to ≤ 45 years at the time of pre-examination
* Volunteer's BMI is ≥ 18.5 and ≤ 29.9
* Volunteer has a stool frequency of at least 3 bowel movements per week
* Volunteer is able and willing to comply with the study instructions
* Volunteer is suitable for participation in the study according to the investigator/study personnel
* Written informed consent is given by volunteer

Exclusion Criteria:

* No command of any local language
* Previously or currently diagnosed neurological or psychiatric disorders
* Previous history of renal, hepatic, cardiovascular disease or clinically significant diabetes
* Gastrointestinal disorders including IBS, IBD or other conditions that might affect the gut environment
* Food allergies or intolerances
* Using drugs (e.g. antibiotics, aspirin, proton pump inhibitors) influencing gastrointestinal function (8 weeks before intervention)
* Use of laxatives and labelled pre-and probiotics in the previous 4 weeks before the beginning of intervention
* Volunteers currently involved or will be involved in another clinical or food study
* History of drug (recreational) or alcohol abuse.
* Use of anti-depressants medication including selective serotonin receptor inhibitors or Amitriptyline for 3 months prior to commencing the trial
* Received bowel preparation for investigative procedures in the 4 weeks prior to the study
* Undergone surgical resection of any part of the bowel.
* pregnant or lactating

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Bifidobacterium spp in stool samples | 4 weeks
  Bifidobacterium spp. will be assessed in stool samples by molecular biological methods
Anxiety with State-Trait Anxiety Inventory questionnaire | 4 weeks
  Anxiety will be assessed with anxiety questionnaire at baseline and at the end of intervention
Depression with Beck's Depression Inventory questionnaire | 4 weeks
  Depression will be assessed with depression questionnaire at baseline and at the end of intervention
Salivary IgA | 4 weeks
  Salivary IgA will be assessed by ELISA at baseline and at the end of intervention

SECONDARY OUTCOMES:
Total bacteria in stool samples | 4 weeks
  Total bacteria will be assessed in stool samples by molecular biological methods
Changes in microbiota composition | 4 weeks
  Microbiota composition at baseline and end will be assessed by 16S rRNA gene sequencing
Stool frequency | 5 weeks
  Stool frequency will be assessed as effective number of bowel movements in a daily diary during baseline and intervention periods
Stool consistency according to Bristol Stool Form Scale | 5 weeks
  Stool consistency will be assessed in a daily diary during baseline and intervention periods
Urinary Metabolites (organic compounds) concentration | 4 weeks
  Urinary Metabolites concentration will be assessed at baseline and end with NMR
Gastrointestinal sensations (bloating) | 5 weeks
  Gastrointestinal sensations (bloating) will be assessed in a daily diary during baseline and intervention periods on a 4-point Likert scale (higher scores indicate higher sensation)
Gastrointestinal sensations (flatulence) | 5 weeks
  Gastrointestinal sensations (flatulence) will be assessed in a daily diary during baseline and intervention periods on a 4-point Likert scale (higher scores indicate higher sensation)
Gastrointestinal sensations (abdominal pain) | 5 weeks
  Gastrointestinal sensations (abdominal pain) will be assessed in a daily diary during baseline and intervention periods on a 4-point Likert scale (higher scores indicate higher sensation)
Gastrointestinal sensations (fullness) | 5 weeks
  Gastrointestinal sensations (fullness) will be assessed in a daily diary during baseline and intervention periods on a 4-point Likert scale (higher scores indicate higher sensation)
Sleep quality via The Pittsburgh Sleep Quality Index | 4 weeks
  Sleep quality will be assessed at baseline and end with The Pittsburgh Sleep Quality Index questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Rastall, Prof, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson PP, Wijeyesekera A, Williams CM, Theis S, van Harsselaar J, Rastall RA. Inulin-type fructans and 2'fucosyllactose alter both microbial composition and appear to alleviate stress-induced mood state in a working population compared to placebo (maltodextrin): the EFFICAD Trial, a randomized, controlled trial. Am J Clin Nutr. 2023 Nov;118(5):938-955. doi: 10.1016/j.ajcnut.2023.08.016. Epub 2023 Aug 30. PMID 37657523